CLINICAL TRIAL: NCT03946696
Title: Bonding at the Very End Emerging Personhood During End-of-life and Palliative Care Through Animal-Assisted Therapy (AAT)
Brief Title: Animal-Assisted Therapy for People With Dementia
Acronym: AATPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Principal Investigator, Cristina Douglas, Postgraduate researcher, University of Aberdeen
Other Study IDs: 2-097-18
Record Dates: First submitted 2018-10-29; First posted 2019-05-13 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Dementia
Keywords: dementia; Animal-Assisted Therapy; ethnography; qualitative study
MeSH Terms: conditions — Dementia | interventions — Drug Interactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dementia: Observations of communication and interactions between people with dementia living in a care home and therapy-animals.
  Interventions: Other: Interactions with therapy-animals

INTERVENTIONS:
Other: Interactions with therapy-animals — How people interact with humans and non-humans animals during and outside visits from therapy-animal teams.

SUMMARY:
This study is a qualitative anthropological research that explores the effects of Animal-Assisted Therapy (AAT) for people with moderate and severe dementia living in a care facility. In particular, the study explores the effects that AAT can have on people with moderate and later stages of dementia, living in a care facility, on: Behavioural and Psychological Symptoms of Dementia (BPSD); mood (depression); quality of life; activity (physical). The AAT effects on people with moderate and later stages of dementia will be compared with effects that other activities provided in the care facility where participants live, may have on the same participants.

This study does not test hypotheses.

DETAILED DESCRIPTION:
This study is a qualitative anthropological research that explores the effects of Animal-Assisted Therapy (AAT) for people with moderate and severe dementia living in a care facility. In particular, the study explores the effects that AAT can have on people with moderate and later stages of dementia, living in a care facility, on: Behavioural and Psychological Symptoms of Dementia (BPSD); mood (depression); quality of life; activity (physical). The AAT effects on people with moderate and later stages of dementia will be compared with effects that other activities provided in the care facility where participants live, may have on the same participants.

AAT is defined as an activity provided by a handler and his/her animal (e.g., dog, cat, rabbit, bird, horse) for somebody living with a certain medical condition/illness. AAT is different than Assistant Dogs/Animal (e.g., guide dogs for the blind), who have a very specific training. In this research, we will focus mostly on therapy-dogs and therapy-owls for people with dementia living in care homes.

The research will be conducted over a period of 12 months. The primary methods that will be used are participant observation (accompanying and observing volunteers during animal-assisted therapy meetings and various activities in the care homes) and interviewing the residents, care homes' staff, volunteers, canine trainers and veterinarians. Additional data will be collected through document analysis (consulting care home policies and participants' care plans and medical notes) and auto-ethnography (auto-observations of interactions between the student and 2 dogs).

The instruments described in the outcome measures are used as guidance only. As this research is non-quantitative, the items listed in the scale instruments are not administered like in a usual clinical testing. The specificity of anthropological research, especially in regard to the use of its methods (participant observation, triangulated with in-depth interview, document analysis and auto-ethnography) addresses implicitly the limitations of such instruments.

While the focus of the research remains on the interactions between people with dementia and therapy-animals, the involvement of the other participants offers different perspectives of looking at these interactions and at their context. For anthropological research, it is fundamental that a certain topic/issue is addressed in its context by gathering information from multiple perspectives. This has been documented as being one of the biggest strengths of anthropological research investigating a clinical-related topic.

The aim of this research is to understand what are the effects that therapy-animals can have on people living with dementia (in moderate and severe stages) in a care facility. While it doesn't aim to compare people living with dementia in their own homes and their potential interaction with a therapy-animal, the research compares the effects of AAT with other activities (e.g., music therapy; craft therapy) and in the context of human interactions (e.g., interactions with other residents; care facility staff members; family members). Because it is documented that animals' therapeutic effects are possible through bond transference, the research also looks as part of the context at how the human-animal bond is formed, how can be transferred and how participants may develop a bond with the therapy-animal. This will be done by interviewing therapy-animal volunteers; canine trainers; and veterinarians. While these might appear as two different projects, we argue that this perspective (how the human-animal bond is formed and its potential therapeutic effect in being transferred) can offer new and original insights in understanding dementia and its stages, as well as a more accurate understanding of AAT effects on people with moderate and severe dementia.

Although the benefits of Animal-Assisted Therapy have been previously documented, these were mostly statistical or experimental studies. To date, there is no study that explores the relationship between therapy-animals and people with dementia using a long-term qualitative approach. Almost all the studies consulted in preparation for our protocol recommend a research that approaches AAT for people with dementia in the context of social interactions and living conditions and from the perspectives described by us. The lack of the context and of these perspectives have been documented/acknowledged as limitations of previous studies in understanding the effects of AAT for people with dementia. These limitations are addressed in our study by looking at them from the diversity of the perspectives we propose.

Given the increased number of people living with dementia, the moral imperative of offering them activities that enhance their quality of life especially in later stages, as well as the rising literature documenting the benefits of companion animals, we aim that this research to contribute to new approaches and policies of care for people with moderate and severe dementia.

ELIGIBILITY:
Inclusion Criteria:

1. People diagnosed with moderate and severe dementia living in a nursing home, age range 55-100.
2. The above-mentioned participants who receive therapy-animal services.

Exclusion Criteria:

1. People with other medical conditions who receive visits from therapy-animals and who do not reside in a care home.
2. People with dementia who do not reside in a care home.
3. People with dementia younger than 55 years old who live in their own home.

Ages: 55 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People with moderate and severe dementia living in a care home; who are visited by therapy-animal teams.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-07-15 (Estimated); Primary Completion 2022-07-14 (Estimated); Study Completion 2023-07-14 (Estimated)

PRIMARY OUTCOMES:
Behavioural and Psychological Symptoms of Dementia (BPSD) | 12 months
  Observations of behaviours associated with dementia (wandering; agitation; anxiety; irritability; apathy; disinhibition). Please note this is a qualitative study that does not use measuring tools.
Symptoms of Depression in dementia | 12 months
  Observation - Please note this is a qualitative study that does not use measuring tools.
Verbal and non-verbal aspects of communication in dementia (e.g., smile; touch; direction of gaze); words. | 12 months
  Observations and interviews - Please note this is a qualitative study that does not use measuring tools.

SECONDARY OUTCOMES:
Patient experience of Animal-Assisted Therapy visits | 15 minutes-1 hour
  Qualitative evaluation of patient experience of visits from a therapy-animal team assessed in qualitative in-depth interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Whitehouse, Principal Investigator — University of Aberdeen
Locations (1):
- University of Aberdeen, Aberdeen, Aberdeenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only the main researcher Cristina Douglas will have access to primary data.